CLINICAL TRIAL: NCT03377842
Title: A Real World Study of Efficacy and Safety for Apatinib Treatment as the Neoadjuvant Therapy in Advanced Colorectal Cancer
Brief Title: Apatinib Treatment as the Neoadjuvant Therapy in Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Zhao gaoping, chief physician, Sichuan Provincial People's Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APTN-CRC-201712
Record Dates: First submitted 2017-12-08; First posted 2017-12-19 (Actual); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Colorectal Cancer; Neoadjuvant Therapy
Keywords: apatinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Folfox protocol; apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFOX regimen (Active Comparator): FOLFOX regime alone.
  Interventions: Drug: FOLFOX regimen
- Apatinib and FOLFOX regimen (Experimental): Apatinib combine with FOLFOX regimen.
  Interventions: Drug: apatinib and FOLFOX regimen

INTERVENTIONS:
Drug: FOLFOX regimen — FOLFOX(Oxaliplatin 85 mg/m² IV infusion and leucovorin 200 mg/m² IV infusion， followed by Fluorouracil 400 mg/m² IV bolus , followed by Fluorouracil 600 mg/m²/h IV infusionas a 22-hour continuous infusion). Repeat cycle every 2 weeks for a total of 6 cycl
  Arms: FOLFOX regimen
Drug: apatinib and FOLFOX regimen — Apatinib, 500mg p.o. qd, Repeat cycle every 2 weeks for a total of 6 cycles. FOLFOX regime, Repeat cycle every 2 weeks for a total of 6 cycles.
  Arms: Apatinib and FOLFOX regimen

SUMMARY:
Apatinib has been proved to be effective and safe among patients in advanced colorectal cancer in several trials. the investigators aimed to evaluate its efficacy and safety as the neoadjuvant therapy in real world practice, and to explore factors associated with efficacy.

DETAILED DESCRIPTION:
Regorafenib (BAY 73-4506, commercial name Stivarga) is an oral multi-kinase inhibitor developed by Bayer which shows anti-angiogenic activity due to its dual targeted VEGFR2-TIE2 tyrosine kinase inhibition.Regorafenib demonstrated to increase the overall survival of patients with metastatic colorectal cancer and has been approved by the CFDA in 2017.

Apatinib, a small molecule receptor tyrosine kinase (RTK) inhibitor, targets the intracellular domain of the VEGFR-2 ATP binding site, and is the first anti-angiogenic therapy approved by the China Food and Drug Administration in December 2014 for the treatment of metastatic gastric cancer in third-line or later treatment. It is an orally bioavailable, small molecule agent which is thought to inhibit angiogenesis in cancer cells; specifically apatinib inhibits VEGF-mediated endothelial cell migration and proliferation thus blocking new blood vessel formation in tumor tissue. It is an investigational cancer drug currently undergoing clinical trials as a potential targeted treatment for metastatic gastric carcinoma, metastatic breast cancer ,advanced hepatocellular carcinoma and advanced colorectal cancer.

Apatinib are often used in advanced colorectal cancer for uses that are not within its approved indication for use.However, the knowledge gained from all uses of apatinib in this medical practice is often not realized because the data collected are not systematically characterized, aggregated, and analyzed in a way that can be relied upon to inform its further usage.

In some cases, a "traditional" clinical trial may be impractical or excessively challenging to conduct. Ethical issues regarding treatment assignment, and other similar challenges, may present themsevels when developing and attempting to execute a high quality clinical trial. Analyses of real-world data(RWD), using appropriate methods, may in some cases provide similar information with comparable or even superior characteristics to information collected and analyzed through a traditional clinical trial. For example, RWD collected using a randomized exposure assignment within a registry can provide a sufficient number of patients for powered subgroup analyses.

the investigators will evaluate the efficacy and safety for Apatinib combine with other chemotherapy regimens as the neoadjuvant therapy in advanced colorectal cancer in a real world study setting. This study leveraging RWD can potentially provide information on a wider patient population, thus providing information that cannot be obtained through a traditional clinical trial alone.

ELIGIBILITY:
Inclusion Criteria:

* Age of 18 years or older.
* Histological or cytological confirmation of adenocarcinoma of the colon or/and rectum;
* Stage TxNxM1 (truly metastatic disease) with liver metastases only.
* Patients should be voluntary to the trial and provide with signed informed consent.
* The researchers believe patients can benefit from the study.

Exclusion Criteria:

* Patients with a known history of allergic reactions and/or hypersensitivity attributed to apatinib or its accessories.
* Pregnant or lactating women
* Patients with Apatinib contraindications
* Patients of doctors considered unsuitable for the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-01-31 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
R0 ,R1 or R2 resection | at least 4-6 weeks after the end of chemotherapy
  Number of patients (%) with hepatic metastases R0 ,R1 or R2 resection.
Progression-free survival (PFS) | 8 months
  Progression-free survival is defined as the time from randomization to progression (RECIST v1.1 criteria) or death. Patients alive without progression will be censored at the last follow-up.

SECONDARY OUTCOMES:
ORR(objective response rate) | after 8 weeks
  The objective response rate (CR and PR) will be evaluated by the investigator with RECIST v1.1 criteria after 4 cycles.
Overall survival (OS) | 14 months
  Overall survival is defined as the time from randomization to death any cause or last follow-up news for patients alive (censored data).

CONTACTS AND LOCATIONS:
Overall Officials: Gaoping Gaoping, doctor, Study Chair — Sichuan province hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li J, Qin S, Xu J, Xiong J, Wu C, Bai Y, Liu W, Tong J, Liu Y, Xu R, Wang Z, Wang Q, Ouyang X, Yang Y, Ba Y, Liang J, Lin X, Luo D, Zheng R, Wang X, Sun G, Wang L, Zheng L, Guo H, Wu J, Xu N, Yang J, Zhang H, Cheng Y, Wang N, Chen L, Fan Z, Sun P, Yu H. Randomized, Double-Blind, Placebo-Controlled Phase III Trial of Apatinib in Patients With Chemotherapy-Refractory Advanced or Metastatic Adenocarcinoma of the Stomach or Gastroesophageal Junction. J Clin Oncol. 2016 May 1;34(13):1448-54. doi: 10.1200/JCO.2015.63.5995. Epub 2016 Feb 16. PMID 26884585
- See also: descriptions about real world study issued by the FDA — https://www.fda.gov/ScienceResearch/SpecialTopics/RealWorldEvidence/default.htm